CLINICAL TRIAL: NCT02861248
Title: Fractional Microplasma Radiofrequency Technology for Non-hypertrophic Post-burn Scars in Asians: A Prospective Study of 95 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, M.D., Ph.D., Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Plasma-1
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Cicatrix
Keywords: Burn Scar; Micro-plasma Radiofrequency Therapy
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser treatment (Experimental): Fractional micro-plasma radiofrequency treatment given to 95 patients with non-hypertrophic burn scar.
  Interventions: Procedure: Fractional micro-plasma radiofrequency treatment

INTERVENTIONS:
Procedure: Fractional micro-plasma radiofrequency treatment — After the patient's scars were subjected to a mild cleanser and 70% alcohol, a topical cream of 5% lidocaine hydrochloric acid (Beijing Ziguang Medication Manufacture Corporation Ltd, Beijing, China) was applied to the entire scar surface under occlusion for 60-90 min before treatment to achieve local anesthesia. Fractional micro-plasma radiofrequency treatment (Pixel RF, Accent XL; Alma Lasers, Caesarea, Israel) was applied using a roller tip at 50-80 watts. Three or four passes were made in different directions over each affected area. A high rolling speed of roughly 5 cm/s was manually controlled. This treatment was accompanied by an air cooler (Cryo 5; Zimmer, Warsaw, IN, USA) for pain control. All patients attended three to five treatment sessions at intervals of 8-16 weeks.

SUMMARY:
A prospective study to evaluate the efficacy and safety of FMRT for treating non-hypertrophic post-burn scars in an Asian population.

DETAILED DESCRIPTION:
Background: Laser therapy is an emerging, minimally invasive treatment for scars. Among the various techniques, fractional microplasma radiofrequency technology (FMRT) has proved to be effective for various types of scars and skin conditions such as rhytids, striae distensae, and hyperpigmentation.

Method: A prospective clinical trial was conducted to evaluate the efficacy and safety of FMRT for treating non-hypertrophic post-burn scars in an Asian population. All patients underwent three to five treatment sessions at intervals of 8-16 weeks. The patient and observer scar assessment scales (POSAS) were use to evaluate changes in the burn scars before and after treatment. Intermediate and long-term adverse events were recorded for outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with ≥1-year-old non-hypertrophic burn scars

Exclusion Criteria:

* pregnancy or breastfeeding
* history of hypertrophic scars or keloids
* abnormal medical examination including routine blood count, liver and kidney functions and immune function
* history of treatment including surgery, dermabrasion, laser treatment within the past 6 months
* the presence of a cardiac pacemaker or other metallic implant near the treatment site.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
POSAS score | From baseline to 6 months after final treatment
  The patient component of the POSAS contains six parameters that the patient scores: pain, itching, color, stiffness, thickness, relief. The physician (observer) component contains five parameters: vascularization, pigmentation, pliability, thickness, relief. Each parameter is scored from 1 to 10, with 1 indicating that the scar similar to normal skin and 10 indicating the worst situation imaginable.

SECONDARY OUTCOMES:
Complications | From baseline to 6 months after final treatment
  Complication including edema, erythema, infection, dyschromia, hypertrophic scar formation or any other complications reported

CONTACTS AND LOCATIONS:
Locations (1):
- Laser division of Plastic Surgery Department, Shanghai 9th people's hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided